CLINICAL TRIAL: NCT00003293
Title: A Phase III Randomized Study of SU101 Versus Procarbazine for Patients With Glioblastoma Multiforme in First Relapse
Brief Title: SU-101 Compared With Procarbazine in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SUGEN-SU101.015; CDR0000066226; MSKCC-98020; UCLA-HSPC-980105201
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Leflunomide; Procarbazine

INTERVENTIONS:
Drug: leflunomide
Drug: procarbazine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether SU-101 is more effective than procarbazine in treating patients with glioblastoma multiforme.

PURPOSE: Randomized phase III trial to compare the effectiveness of SU-101 with that of procarbazine in treating patients with glioblastoma multiforme that has recurred.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the median survival of patients with glioblastoma multiforme in first relapse treated with intravenous leflunomide (SU101) administered as a loading dose with weekly maintenance therapy versus oral, single-agent procarbazine administered daily for 28 days every 56 days. II. Compare the median time to progression for these regimens in these patients. III. Assess the objective response of these patients. IV. Assess the safety of SU101 given on this schedule. V. Describe the health-related quality of life of these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to performance status (Karnofsky 60-80% vs 90-100%), age (less than 50 vs 50 and over), and time from initial diagnosis to recurrence (6 months or greater vs less than 6 months). Patients are randomized to one of two treatment arms. Arm I: Patients receive leflunomide (SU101) IV over 6 hours daily on days 1-4, again 4-8 days later, and weekly thereafter for a total of 4 loading dose infusions and six maintenance infusions in course 1. Patients receive 7 weekly maintenance infusions of SU101 in courses thereafter. Treatment repeats every 8 weeks. Arm II: Patients receive procarbazine orally once or twice daily for 4 weeks. Treatment is repeated every 8 weeks. All patients complete a health-related quality-of-life questionnaire every 8 weeks and at study withdrawal. Treatment courses continue up to a maximum of 1 year in the absence of unacceptable toxicity or disease progression. Patients are followed every 2 months, beginning 30 days after study completion.

PROJECTED ACCRUAL: A maximum of 380 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven refractory or recurrent supratentorial glioblastoma multiforme Bidimensionally measurable, enhancing residual disease by T1-weighted gadolinium-enhanced MRI required within 15 days prior to treatment Stable dose of corticosteroids required for at least 7 days prior to scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 9 g/dL without blood transfusions for 15 days prior to treatment Hepatic: AST/SGOT no greater than 3 times upper limit of normal (ULN) Bilirubin less than 1.5 times ULN Renal: Creatinine no greater than 2 mg/dL OR Creatinine clearance at least 40 mL/min Other: Not allergic to etoposide Effective contraception required of fertile patients Negative serum pregnancy test required of fertile women No other acute or chronic medical or psychiatric condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior leflunomide (SU101) therapy No more than one prior single-agent or combination systemic chemotherapy regimen for initial disease Radiosensitizer(s) concurrent with radiotherapy allowed in addition to chemotherapy for primary disease At least 6 weeks since nitrosourea or mitomycin At least 2 weeks since vincristine No prior single-agent procarbazine At least 4 weeks since other chemotherapy No concurrent chemotherapy agents Endocrine therapy: No concurrent hormone therapy (except medroxyprogesterone acetate for appetite stimulation) Less than 4 weeks of prior hormonal therapy (tamoxifen or retinoids) if failed one prior chemotherapy regimen Radiotherapy: Prior conventional radiotherapy for initial disease required No more than one prior course of radiotherapy At least 8 weeks since radiotherapy No prior interstitial radiotherapy No concurrent radiotherapy Surgery: Maximally feasible resection for initial disease required No more than two resections permitted At least 1 week since surgery and/or biopsy for disease No prior interstitial radiotherapy or implanted BCNU-wafers No concurrent surgery (including resection, stereotactic surgery or interstitial implants) Other: No concurrent investigational agent At least 4 weeks since prior investigational agent At least 1 week since cholestyramine or monoamine oxidase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison L. Hannah, MBBS, Study Chair — SUGEN
Locations (35):
- United States (32):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - St. Francis Hospital, San Francisco, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Medical College of Georgia Hospital and Clinics, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Center of Albany Medical Center, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario